CLINICAL TRIAL: NCT03666741
Title: Clinical Outcomes of Patients Under the Age of Sixty Undergoing INSPIRIS RESILIA Aortic Valve Replacement
Brief Title: Inspiris Resilia Durability Registry
Acronym: INDURE
Status: Active, not recruiting | Type: Observational
Sponsor: Institut für Pharmakologie und Präventive Medizin (Network)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: HVT-R18-IND
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Aortic Valve Stenosis
Keywords: Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases; Surgical valve
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | US Export: No

INTERVENTIONS:
Device: AVR with or without CABG — Surgical aortic valve implantation with INSPIRIS RESILIA Aortic Valve™

SUMMARY:
Prospective, open-label, multicenter, European registry with a follow-up of 5 years to assess the clinical outcomes of patients younger than 60 years who undergo surgical AVR with the INSPIRIS RESILIA Aortic Valve™.

DETAILED DESCRIPTION:
The INSPIRIS RESILIA Aortic Valve™ is a stented tri-leaflet valve comprised of bovine pericardial tissue. The tissue is created by treating bovine pericardial tissue with Edwards Integrity Preservation. It incorporates a stable capping anticalcification process, which blocks residual aldehyde groups known to bind with calcium. Tissue preservation with glycerol allows the valve to be stored without a traditional liquid-based solution, such as glutaraldehyde. Therefore, valve is stored under dry packaging conditions and consequently does not require rinsing prior to implantation.

The novel tissue preservation technology significantly improves hemodynamic and anticalcification properties compared with the standard Perimount valve in an ovine model. In this registry, data is collected over a period of 5 years to demonstrate these properties in a clinical real-life setting. Clinical outcomes, hemodynamic as well as safety parameters and quality of life data are documented into e-CRF at baseline, surgery, pre-discharge, 3-6 months and annually up to year 5.

The required sample size was calculated using the online calculator at http://www.surveysystem.com/sscalc.htm. It was estimated, from COMMENCE Trial dataset that freedom from time-related valve safety events at 1 year (composite endpoint according to VARC-2) is around 0.915. The following table illustrates 95% CIs at different levels of risk:

Sample Size Observed freedom from event 95%CI 400 0.900 ± 0.0294 400 0.910 ± 0.0280 400 0.915 ± 0.0214 400 0.920 ± 0.0266 400 0.930 ± 0.0250

20% of registry sites will be monitored with 100% source data verification

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 60 years inclusive
2. Subject requiring a planned replacement of their native aortic valve as indicated in a preoperative evaluation
3. Subject is scheduled to undergo planned aortic valve replacement with or without concomitant root replacement and/or coronary bypass surgery
4. Subject is scheduled to attend yearly follow-up visits at the registry center up to 5 years follow-up
5. Subject provides written informed consent prior to the procedure

Exclusion Criteria:

1. Active endocarditis/myocarditis or endocarditis/myocarditis within 3 months prior to the scheduled aortic valve replacement surgery
2. Previous aortic valve replacement
3. Valve implantation is not possible in accordance with the device IFU
4. Subject has a life expectancy ≤ 12 months for any reason

Intraoperative Exclusion criteria:

1. Valve implantation is not possible in accordance with the device IFU

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients under the age of 60 with an indication for surgical AVR who will receive an Edwards INSPIRIS RESILIA aortic valve prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Time-related valve safety | Year 1
  Composite endpoint according to VARC-2 depicted as freedom from event:
  * SVD (structural valve deterioration)
  * Valve-related dysfunction
  * Requirement of repeat procedure
  * Prosthetic valve endocarditis
  * Prosthetic valve thrombosis
  * Thromboembolic events (e.g. stroke)
  * Valve-related VARC bleeding
Freedom from severe SVD (structural valve deterioration) | Year 5
  Freedom from stage 3 SVD including stenosis and regurgitation determined by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bramlage, Professor, Study Director — CEO IPPMed; Ruggero dePaulis, Professor, Principal Investigator — European Hospital Rome, Italy; Bart Meuris, Professor, Principal Investigator — UZ Leuven, Belgium
Locations (21):
- Austria (3):
  - University Clinics St. Pölten, Sankt Pölten
  - Heart Center Hietzing, Vienna
  - Medical University Vienna, Vienna
- KU Leuven, Leuven, Belgium
- Canada (2):
  - Institut de Cardiologie de Montréal, Université de Montréal, Montreal
  - Laval University, Québec
- France (4):
  - Hopital de la Timone, Marseille
  - L'institut du thorax - CHU (Centre Hospitalier Universitaire de Nantes), Nantes
  - Centre Hospitalier Universitaire (CHU) de Rennes, Rennes
  - CHRU - Hospital Trousseau, Tours
- Germany (2):
  - UNIVERSITÄTSKLINIKUM FREIBURG, Universitäts-Herzzentrum Herz- und Gefäßchirurgie, Freiburg im Breisgau, Baden-Wurttemberg
  - Heart Center Leipzig, Leipzig
- Italy (4):
  - University Hospital Careggi, Florence
  - Centro Cardiologico Monzino, Milan
  - European Hospital Rome, Roma
  - AOU San Giovanni di Dio e Ruggi d'Aragona, Salerno
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- University Hospital Virgen de la Arrixaca, Murcia, Spain
- United Kingdom (3):
  - NHS Lothian, Edinburgh
  - Glenfield Hospital, Glenfield
  - King's College Hospital NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Flameng W, Hermans H, Verbeken E, Meuris B. A randomized assessment of an advanced tissue preservation technology in the juvenile sheep model. J Thorac Cardiovasc Surg. 2015 Jan;149(1):340-5. doi: 10.1016/j.jtcvs.2014.09.062. Epub 2014 Sep 28. PMID 25439467
- [Background] Puskas JD, Bavaria JE, Svensson LG, Blackstone EH, Griffith B, Gammie JS, Heimansohn DA, Sadowski J, Bartus K, Johnston DR, Rozanski J, Rosengart T, Girardi LN, Klodell CT, Mumtaz MA, Takayama H, Halkos M, Starnes V, Boateng P, Timek TA, Ryan W, Omer S, Smith CR; COMMENCE Trial Investigators. The COMMENCE trial: 2-year outcomes with an aortic bioprosthesis with RESILIA tissue. Eur J Cardiothorac Surg. 2017 Sep 1;52(3):432-439. doi: 10.1093/ejcts/ezx158. PMID 28605428
- [Background] Kappetein AP, Head SJ, Genereux P, Piazza N, van Mieghem NM, Blackstone EH, Brott TG, Cohen DJ, Cutlip DE, van Es GA, Hahn RT, Kirtane AJ, Krucoff MW, Kodali S, Mack MJ, Mehran R, Rodes-Cabau J, Vranckx P, Webb JG, Windecker S, Serruys PW, Leon MB; Valve Academic Research Consortium-2. Updated standardized endpoint definitions for transcatheter aortic valve implantation: the Valve Academic Research Consortium-2 consensus document. EuroIntervention. 2012 Nov 22;8(7):782-95. doi: 10.4244/EIJV8I7A121. PMID 23022744
- [Background] Dvir D, Bourguignon T, Otto CM, Hahn RT, Rosenhek R, Webb JG, Treede H, Sarano ME, Feldman T, Wijeysundera HC, Topilsky Y, Aupart M, Reardon MJ, Mackensen GB, Szeto WY, Kornowski R, Gammie JS, Yoganathan AP, Arbel Y, Borger MA, Simonato M, Reisman M, Makkar RR, Abizaid A, McCabe JM, Dahle G, Aldea GS, Leipsic J, Pibarot P, Moat NE, Mack MJ, Kappetein AP, Leon MB; VIVID (Valve in Valve International Data) Investigators. Standardized Definition of Structural Valve Degeneration for Surgical and Transcatheter Bioprosthetic Aortic Valves. Circulation. 2018 Jan 23;137(4):388-399. doi: 10.1161/CIRCULATIONAHA.117.030729. PMID 29358344
- [Background] Capodanno D, Petronio AS, Prendergast B, Eltchaninoff H, Vahanian A, Modine T, Lancellotti P, Sondergaard L, Ludman PF, Tamburino C, Piazza N, Hancock J, Mehilli J, Byrne RA, Baumbach A, Kappetein AP, Windecker S, Bax J, Haude M. Standardized definitions of structural deterioration and valve failure in assessing long-term durability of transcatheter and surgical aortic bioprosthetic valves: a consensus statement from the European Association of Percutaneous Cardiovascular Interventions (EAPCI) endorsed by the European Society of Cardiology (ESC) and the European Association for Cardio-Thoracic Surgery (EACTS). Eur J Cardiothorac Surg. 2017 Sep 1;52(3):408-417. doi: 10.1093/ejcts/ezx244. No abstract available. PMID 28874031
- [Derived] De Paulis R, Bakhtiary F, Ahmad AE, Andreas M, Autschbach R, Benedikt P, Binder K, Bonaros N, Borger M, Bourguignon T, Canovas S, Coscioni E, Dagenais F, Demers P, Dewald O, Doll N, Feyrer R, Geissler HJ, Grabenwoger M, Grunenfelder J, Kueri S, Lam KY, Langanay T, Laufer G, Van Leeuwen W, Karimli S, Liebold A, Mariscalco G, Massoudy P, Mehdiani A, Pessotto R, Pollari F, Poling J, Polvani G, Ricci A, Roussel JC, Salamate S, Siepe M, Stefano P, Strauch J, Theron A, Votsch A, Weber A, Wendler O, Thielmann M, Eden M, Botta B, Bramlage P, Meuris B, Zierer A. Gender-based outcomes following surgical aortic valve replacement: a multicentre propensity score matching analysisdagger. Eur J Cardiothorac Surg. 2025 Jul 1;67(7):ezaf099. doi: 10.1093/ejcts/ezaf099. PMID 40608978
- [Derived] Meuris B, Roussel JC, Borger MA, Siepe M, Stefano P, Laufer G, Langanay T, Theron A, Grabenwoger M, Binder K, Demers P, Pessotto R, van Leeuwen W, Bourguignon T, Canovas S, Mariscalco G, Coscioni E, Dagenais F, Wendler O, Polvani G, Eden M, Botta B, Bramlage P, De Paulis R. Durability of bioprosthetic aortic valve replacement in patients under the age of 60 years - 1-year follow-up from the prospective INDURE registry. Interdiscip Cardiovasc Thorac Surg. 2023 Oct 4;37(4):ivad115. doi: 10.1093/icvts/ivad115. PMID 37462612
- [Derived] Meuris B, Borger MA, Bourguignon T, Siepe M, Grabenwoger M, Laufer G, Binder K, Polvani G, Stefano P, Coscioni E, van Leeuwen W, Demers P, Dagenais F, Canovas S, Theron A, Langanay T, Roussel JC, Wendler O, Mariscalco G, Pessotto R, Botta B, Bramlage P, de Paulis R. Durability of bioprosthetic aortic valves in patients under the age of 60 years - rationale and design of the international INDURE registry. J Cardiothorac Surg. 2020 May 27;15(1):119. doi: 10.1186/s13019-020-01155-6. PMID 32460798